CLINICAL TRIAL: NCT03262857
Title: Comparison of the Success Rate of Anesthesia Between Lidocaine 2% and Lidocaine 2% Mixed With 10% Magnesium Sulfate in the Inferior Alveolar Nerve Block in Posterior Teeth With Irreversible Pulpitis
Brief Title: Effect of Lidocaine With Magnesium Sulfate on the Success of the Inferior Alveolar Nerve Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Amir Mousavi, Assistant Professor of Endodontics, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUMS 396169
Record Dates: First submitted 2017-08-19; First posted 2017-08-25 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Local Anesthesia
Keywords: magnesium sulfate; pulpitis; anesthesia
MeSH Terms: conditions — Pulpitis | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- time of start of anesthesia (Experimental)
  Interventions: Drug: use of magnesium sulfate with lidocaine in inferior alveolar nerve block
- intensity of anesthesia (Experimental)
  Interventions: Drug: use of magnesium sulfate with lidocaine in inferior alveolar nerve block

INTERVENTIONS:
Drug: use of magnesium sulfate with lidocaine in inferior alveolar nerve block

SUMMARY:
68 healthy patients pulpitis and requiring root canal therapy are selected. . Sampling was done in a simple and non-experimental way from a dental clinic in Isfahan, and then the samples were randomly assigned to one of the two experimental groups (A, B) using simple random numbers.

Each vial is filled with distilled water or magnesium sulfate by an individual who is unaware of the nature of the design and is not involved in the design, and each letter A or B is written. This statement is not decoded after the statistical examination. Therefore, the study is blind and blind. In this way, 60 patients are examined in 2 groups of 34 First, patients with recognized pulpitis in mandibular posterior teeth have been identified and information about them is given. Patients will be introduced to the executive phase after the required explanation and clarification of the ambiguity and written consent. After completing the patient information form by the practitioner and complying with all entry and exit criteria, the study begins on each patient.

The patient records his pain as an initial pain on the Heath-Parker Visual Analogue Scale (VAS). This pain measurement method involves a 180 mm line with descriptive words that differentiates patients on a line where the best describes their pain. In order to design a standard injection of the maxillary nerve block in all patients, using Aspirating Dental Injection Syringe, Novocol Ontario, Canada, the needle of the 27 mm long 35 mm (Septoject, Septodont, Saint-Maur-des- Fosses cedex, France) Lidocaine 2% with epinephrine 80000/1 mixed with magnesium sulfate or distilled water, injections in the retro-cell region and cm1 above the occlusal mandibular plan. After insertion of the needle at a rate of 3-5 mm into the tissue, aspiration was performed and about 2-3 ml / 2. It is injected from the contents of the cartridge, the syringe 1 mm is returned to the bone hard tissue (in the form of the syringe body in the perimmel area of the opposite side), and after the aspiration of the contents of each cartridge in a 1 minute period It is injected. After 15 minutes, in case of numbness of the lips, the patient begins to study and the access cavity begins on the desired tooth. In each of the stages of acquiring the access cavity or entering the initial file to the canal, in the event of pain, the treatment is suspended and the patient signs his pain on the pain assessment chart based on the Heft-parker VAS and at this stage the study It's over. In the absence of anesthetized lips, the patient is excluded from the study and after completing the injection, the root canal is given.

DETAILED DESCRIPTION:
68 healthy patients (ASA I, II, and over the age of 18 and under the age of 60 years with posterior mandibular maxillary jaw and with symptomatic pulpitis (severe and long response to cold test) and requiring root canal therapy are selected. .

The criteria for entering the study include: absence of periodontal disease and any periapical radiolucency except for PDL dilation, absence of susceptibility to local anesthetic or sulfite drugs, non-pregnant women and non-lactating women, lack of drugs that interact with local anesthetic Or change the perception of pain (such as beta-blocker drugs, opiates, etc.).

Exclusion criteria included: Clinical observation of necrotic pulp after opening the access cavity in the desired tooth, the patient's inability to give informed consent and patient's continuation of the research in each stage of the trial.

Sampling was done in a simple and non-experimental way from a dental clinic in Isfahan, and then the samples were randomly assigned to one of the two experimental groups (A, B) using simple random numbers.

Preparation of infiltration solution will be such that using a syringe with a high accuracy (hamilton) of 0.2 ml of magnesium 10% sulfate vial or distilled water sterilized and then into a 1.8ml cartridge of lidocaine 2% With an epinephrine 80000/1, the solution is shaken 5 times for mixing, so that no sediment should be seen.

Each vial is filled with distilled water or magnesium sulfate by an individual who is unaware of the nature of the design and is not involved in the design, and each letter A or B is written. This statement is not decoded after the statistical examination. Therefore, the study is blind and blind. In this way, 68 patients are examined in 2 groups of 34 people. It should be noted that all anesthesia is injected by one person.

First, patients with recognized pulpitis in mandibular posterior teeth have been identified and information about them is given. Patients will be introduced to the executive phase after the required explanation and clarification of the ambiguity and written consent. After completing the patient information form by the practitioner and complying with all entry and exit criteria, the study begins on each patient.

The patient records his pain as an initial pain on the Heath-Parker Visual Analogue Scale (VAS). This pain measurement method involves a 180 mm line with descriptive words that differentiates patients on a line where the best describes their pain. In order to design a standard injection of the maxillary nerve block in all patients, using Aspirating Dental Injection Syringe, Novocol Ontario, Canada, the needle of the 27 mm long 35 mm (Septoject, Septodont, Saint-Maur-des- Fosses cedex, France) Lidocaine 2% with epinephrine 80000/1 mixed with magnesium sulfate or distilled water, injections in the retro-cell region and cm1 above the occlusal mandibular plan. After insertion of the needle at a rate of 3-5 mm into the tissue, aspiration was performed and about 2-3 ml / 2. It is injected from the contents of the cartridge, the syringe 1 mm is returned to the bone hard tissue (in the form of the syringe body in the perimmel area of the opposite side), and after the aspiration of the contents of each cartridge in a 1 minute period It is injected. After 15 minutes, in case of numbness of the lips, the patient begins to study and the access cavity begins on the desired tooth. In each of the stages of acquiring the access cavity or entering the initial file to the canal, in the event of pain, the treatment is suspended and the patient signs his pain on the pain assessment chart based on the Heft-parker VAS and at this stage the study It's over. In the absence of anesthetized lips, the patient is excluded from the study and after completing the injection, the root canal is given.

ELIGIBILITY:
Inclusion Criteria:

* absence of periodontal disease
* absence of susceptibility to local anesthetics or sulfite
* non-pregnant women and non-lactating women

Exclusion Criteria:

* Clinical observation of necrotic pulp
* the patient's inability to give informed consent and patient's continuation of the research in each stage of the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Effect of Magnesium with lidocaine | 10 to 20 minute
  measuring the time of starting of anesthesia with questionnaire
intensity of pain | 10-20 minute
  measuring pain after access cavity preparation with questionnaire